CLINICAL TRIAL: NCT05535465
Title: Malaria Control : Improving Access to Prevention, Diagnostic and Care for Vulnerable Rural Communities
Acronym: REACT-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Institut Pierre Richet (Other Government); Expertise France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRD-2-002
Record Dates: First submitted 2022-08-24; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Cluster randomized - Step-wedged design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Heath system strengthening with additional trained mobile health care worker to help community health workers
  Interventions: Other: Public health intervention
- Standard of care (No Intervention): National strategy to control malaria

INTERVENTIONS:
Other: Public health intervention — additional trained mobile health workers are hired to support and supervise the activities of community health workers
  Arms: Intervention arm

SUMMARY:
In the REACT 2 project, a consortium proposes to study in Burkina Faso and Côte d'Ivoire, the impact of a public health intervention in rural communities in order to improve access to malaria therapeutic and preventive arsenal for vulnerable populations (i.e. children, adolescents and pregnant women). The intervention relies on the implementation of mobile health workers to support community health workers.

ELIGIBILITY:
Inclusion Criteria:

* global population

Exclusion Criteria:

* absence of informed consent

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference of malaria incidence between control and intervention arms | Day 0 (cross-sectional survey)
  Incidence will be calculated as the number of malaria cases detected during the cross-sectionnal surveys relative to the population size

SECONDARY OUTCOMES:
Difference of malaria prevalence between control and intervention arms | Day 0 (cross-sectional survey)
  Prevalence will be calculated as the proportion of participants with malaria infection (i.e. positive blood smears) detected during the cross-sectionnal surveys

CONTACTS AND LOCATIONS:
Locations (2):
- IRSS, Bobo-Dioulasso, Houet, Burkina Faso
- IPR, Bouaké, Côte d’Ivoire